## Implementing and Evaluating a Wellness and Social-Emotional Learning Program for Refugee Children During the COVID-19 Pandemic: EMPOWER

# (<u>Em</u>otions <u>Program Outside the Clinic and <u>Wellness Education</u> for <u>Refugees</u>)</u>

ClinicalTrials.gov Identifier: NCT04931888 Documents Last Updated July 20, 2022 Documents Compiled July 23, 2023

| ENGLISH PARENT CONSENT | 2 |
|---------------------------|----|
| ENGLISH ADOLESCENT ASSENT | 7 |
| ENGLISH CHILD ASSENT | 11 |
| DARI PARENT CONSENT | 13 |
| DARI ADOLESCENT ASSENT | 20 |
| DARI CHILD ASSENT | 24 |
| PASHTO PARENT CONSENT | 26 |
| PASHTO ADOLESCENT ASSENT | 31 |
| PASHTO CHILD ASSENT | 35 |

#### ENGLISH PARENT CONSENT

## COMPOUND AUTHORIZATION AND PARENTAL PERMISSION FOR PARTICIPATION IN A RESEARCH STUDY

#### YALE UNIVERSITY SCHOOL OF MEDICINE

<u>Study Title:</u> Implementing and Evaluating a Wellness and Social-Emotional Learning Program for Refugee Children During the COVID-19 Pandemic: EMPOWER

(Emotions Program Outside the Clinic and Wellness Education for Refugees)

<u>Principal Investigator (the person who is responsible for this research):</u> Julia Rosenberg MD MHS 333 Cedar St New Haven. CT

Phone Number: 8609301702

The Academic Pediatric Association, the National Institutes of Health/ National Center of Advancing Translational Science (NIH/NCATS), and Yale University are paying for this study.

#### **Research Study Summary:**

- We are asking you and your child to join a research study.
- The purpose of this research study is evaluate the program that your family will be participating in or has participated in, known as EMPOWER. Evaluations occur before, during, and after participation.
- Study procedures will include: Participation in the program, which your child/children can
  participate in whether or not you decide to be a part of the study. The program will be no different
  for those who do or do not choose to participate in the research study. The study will also include
  answering questions about your and your family's experience in the program and about social and
  emotional health over Zoom.
- Two Zoom surveys are required along with involvement in the summer program (which you can continue regardless of your decision to be a part of the study).
- Participation in the program is also part of this study.
- The zoom surveys will take 2 hours total. The program will involve about 3 person of in-person and 1 hour of zoom activities per week over two weeks.
- There are some risks from participating in this study. Risks include challenges attending in-person activities or not liking in-person activities, and/or discomfort with some of the questions asked.
- The study may have no benefits to your child. The study may benefit others who are interested in learning more about implementing programs similar to EMPOWER.
- There are other choices available to your child outside of this research. Your child does not have to participate in this research even if you are participating in EMPOWER.
- Giving permission for you and your child to take part in this study is your choice. You can choose
  to give permission, or you can choose not to. You can also change your mind at any time.
  Whatever choice you make, your child will not lose access to his or her medical care or give up
  any legal rights or benefits.
- If you are interested in learning more about the study, please continue reading, or have someone
  read to you, the rest of this document. Take as much time as you need before you make your
  decision. Ask the study staff questions about anything you do not understand. Once you
  understand the study, we will ask you if you wish to give permission for your child to participate; if
  so, you will have tell us verbally that you agree

#### Why is this study being offered to my child?

We are asking your child to take part in a research study because your child is participating in the EMPOWER program. We are looking for 30 families and 75 children to be part of this research study including participation in the program and evaluation before and after the program.

#### Who is paying for the study?

The Academic Pediatric Association, the National Institutes of Health/ National Center of Advancing Translational Science (NIH/NCATS), and Yale University are paying for this study.

#### Who is providing other support for the study?

Elena's Light is providing support for this study.

#### What is the study about?

The purpose of this study is to implement and evaluate the program that your family will be participating in or has participated in, known as EMPOWER.

#### What are you asking my child to do and how long will it take?

If you give permission for your child to take part in this study, this is what will happen: we will ask them questions over Zoom, which are similar to the questions we are asking you, at two different time points. We think that the study will take a total of two hours of your and your children's time (combined). This is in addition to participation in the program, which will involve about 3 hours of in person and 1 hour of zoom activity per week over two weeks. We will ask you questions about your experience with the program and will ask you and your children questions about social and emotional health. Some of these questions will be asked more than once.

#### What are the risks and discomforts of participating?

If you and/or your children decide to take part in this study, you and/or your children may experience challenges attending in-person activities or not liking in-person activities, and/or discomfort with some of the questions asked.

There is the possible risk of loss of confidentiality.

#### How will I know about new risks or important information about the study?

We will tell you if we learn any new information that could change your mind about your child taking part in this study.

#### How can the study possibly benefit my child?

Your child **may or may not** benefit from taking part in this study, by learning about health and wellness through the EMPOWER program.

#### How can the study possibly benefit other people?

The benefits to science and other people may include a better understanding of **the benefits of the EMPOWER** program and how to share this program with others.

#### Are there any costs to participation?

You will not have to pay for your child taking part in this study. The only costs include transportation and their coming to the EMPOWER program and zoom interviews.

#### Will my child be paid for participation?

Your child will not be paid for taking part in this study, but you will be paid a \$25 gift card for each instance of you (along with your child) participating in the zoom survey.

#### What are our choices if I decide not to give permission for my child to take part in this study?

Instead of participating in this study, you have some other choices.

Your child could:

- Participate in EMPOWER without being in a study.
- Take part in another study.

#### How will you keep my child's data safe and private?

We will keep information we collect about your child confidential. We will share it with others if you agree to it or when we have to do it because U.S. or State law requires it. For example, we will tell somebody if we learn that someone is hurting a child or an older person.

Your child's information will be deidentified, meaning we will not keep the name of your child along with his or her responses. Instead, there will be a number associated with your and your child's responses. A list connecting numbers and names will be kept on a password protected computer and will be destroyed after the study is completed.

When we publish the results of the research or talk about it in conferences, we will not use your child's name. If we want to use their name, we would ask you both for your permission.

We will also share information about your child with other researchers for future research but we will not use his or her name or other identifiers. We will not ask you for any additional permission.

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. The researchers with this Certificate may not disclose or use information, documents, or biospecimens that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence, for example, if there is a court subpoena, unless you have consented for this use. Information, documents, or biospecimens protected by this Certificate cannot be disclosed to anyone else who is not connected with the research except, if there is a federal, state, or local law that requires disclosure (such as to report child abuse or communicable diseases but not for federal, state, or local civil, criminal, administrative, legislative, or other proceedings, see below); if you have consented to the disclosure, including for your medical treatment; or if it is used for other scientific research, as allowed by federal regulations protecting research subjects.

The Certificate of Confidentiality will not be used to prevent disclosure as required by federal, state, or local law of child abuse and neglect, or harm to self or others.

#### What information will you collect about my child in this study?

The information we are asking to use and share is called "Protected Health Information." It is protected by a federal law called the Privacy Rule of the Health Insurance Portability and Accountability Act (HIPAA). In general, we cannot use or share your child's health information for research without your permission. If you want, we can give you more information about the Privacy Rule. Also, if you have any questions about the Privacy Rule and your rights, you can speak to Yale Privacy Officer at 203-432-5919.

The specific information about your child and their health that we will collect, use, and share includes:

- Research study records without names, which will include responses to survey questions. These survey questions include questions about stress, quality of life, behavioral health, and COVID-19 knowledge.
- Records about phone calls made as part of this research
- Records about your child's attendance at EMPOWER programs

#### How will you use and share my child's information?

We will use your child's information to conduct the study described in this consent form. We may share your child's information with:

• The U.S. Department of Health and Human Services (DHHS) agencies

- Representatives from Yale University, the Yale Human Research Protection Program and the Institutional Review Board (the committee that reviews, approves, and monitors research on human participants), who are responsible for ensuring research compliance. These individuals are required to keep all information confidential.
- Health care providers who provide services to your child in connection with this study.
- The study's Principal Investigator
- Co-Investigators and other investigators
- Study Coordinator and Members of the Research Team
- Data and Safety Monitoring Boards and others authorized to monitor the conduct of the Study

We will do our best to make sure your child's information stays private. But, if we share information with people who do not have to follow the Privacy Rule, your child's information will no longer be protected by the Privacy Rule. Let us know if you have questions about this. However, to better protect your child's health information, agreements are in place with these individuals and/or companies that require that they keep your child's information confidential.

#### Why must I agree to the information in this document?

By agreeing to the information in this form, you will allow researchers to use and disclose your child's information described above for this research study. This is to ensure that the information related to this research is available to all parties who may need it for research purposes. You always have the right to review and copy your child's health information in their medical record.

#### What if I change my mind?

The authorization to use and disclose your child's health information collected during their participation in this study will never expire. However, you may withdraw or take away your permission at any time. You may withdraw your permission by telling the study staff or by writing to *Julia Rosenberg*, 333 *Cedar Street*, *New Haven* at the Yale University, New Haven, CT 06520.

If you withdraw your permission, your child will not be able to stay in this study but the care they get from their doctor outside this study will not change. No new health information identifying your child will be gathered after the date you withdraw your permission. Information that has already been collected may still be used and given to others until the end of the research study to insure the integrity of the study and/or study oversight.

#### What if I want to refuse or end my child's participation before the study is over?

Allowing your child to take part in this study is your choice. You can choose to give permission, or you can choose not to give permission. You also can change your mind at any time. Whatever choice you make, your child will not lose access to his or her medical care or give up any legal rights or benefits.

Your child will be asked to give their assent to be in the study. If they decide they do not want to be in the study, they will not be enrolled in the study even if you have given permission. You will not be told the reason why your child didn't want to participate.

We would still treat your child with standard therapy or, at your request, refer you to a clinic or doctor who can offer this treatment. Not participating or withdrawing later will not harm your child's relationship with their own doctors or with this institution.

To withdraw from the study, you can call a member of the research team at any time and tell them that you no longer want your child to take part.

The researchers may withdraw your child from participating in the research if necessary. **Such as if your child indicates they no longer want to participate.** 

## What will happen with my child's data if they stop participating?

Your child can continue to participate in EMPOWER activities as much or as little as you would like if they stop participating in the Zoom questions. You may request that the data be withdrawn from the research once it is collected.

#### Who should I contact if I have questions?

Please feel free to ask about anything you don't understand.

If you have questions later or if you have a research-related problem, you can call the Principal Investigator at **860-930-1702** 

If you have questions about your child's rights as a research participant, or you have complaints about this research, you call the Yale Institutional Review Boards at (203) 785-4688 or email <a href="mailto:hrpp@yale.edu">hrpp@yale.edu</a>.

#### **Authorization and Permission**

Your verbal agreement which we will document now indicates that you have listened this consent document and that you give permission for your child to be in this study.

We will provide you a copy of this document.

#### ENGLISH ADOLESCENT ASSENT

#### ADOLESCENT ASSENT FOR PARTICIPATION IN A RESEARCH STUDY

#### YALE UNIVERSITY

Study Title: Implementing and Evaluating a Wellness and Social-Emotional Learning Program for Refugee Children During the COVID-19 Pandemic: EMPOWER

(Emotions Program Outside the Clinic and Wellness Education for Refugees)

Principal Investigator (the person who is responsible for this research): Julia Rosenberg, MD

MHS, 333 Cedar St, New Haven, CT

**Phone Number**: 860-930-1702

## Why am I here?

- We are asking you to join a research study.
- The study will look at your experience with the summer program.
- It will take about one hour on two separate occasions, with questions asked on Zoom.
- It will also involve participating in EMPOWER summer program, with about 3 hours in-person and 1 hour on Zoom each week for two weeks.
- This assent form explains the research study and your part in the study.
- Please read it carefully. Take as much time as you need.
- Please ask the study staff questions about anything you do not understand.
- You can ask guestions now or anytime during the study.
- If you join the study, you can change your mind later.
- You can guit the study at any time.
- We will also ask your parents to allow you to be in the study.

#### Why is this study being offered to me?

We are asking you to join a research study because you and your family are participating in a summer program. We are looking for children who participated in the program, and about 70 total people to be part of this study to learn more about what the program is like for you and your family.

#### What is the study about?

The purpose of this study is to evaluate the program that your family will be participating in or has participated in, known as EMPOWER.

#### What will happen during the study?

If you agree to take part in this study, this is what will happen: you will answer questions during two separate interviews on zoom. We will ask you questions about feelings and emotions. You will also be participating in the summer program, which will involve playing games, completing art projects, and learning about health and wellness, and learning about COVID-19 safety and emotions.

## How long will I be in the study?

You will have 2 Zoom visits that will take about 1 hour each. This is in addition to the program, which will be about 3 hours of in-person over two weeks and 1 hour of Zoom per week over four weeks.

#### What are the possible risks of the study?

You may experience some discomfort with some of the questions we ask, meaning that they may be difficult to answer or it may be hard to think about and talk about emotions and feelings. Risks may also include not enjoying or liking the program.

#### How will I learn any new important information about the study?

We will tell you and your parents if we learn any new information that could change your mind about taking part in this study.

## How can the study possibly benefit me or other people?

The study might benefit you by the experiences you will have in the summer program, including learning new games and exercises, and learning about feelings and emotions.

The study might help other people by helping us understand more about the EMPOWER program and how people who participate in the program feel about it.

#### Will it cost any money for me to be in the study?

You will not have to pay for taking part in this study. The only costs include transportation to the program.

#### Will I be paid if I join the study?

You will not be paid for taking part in this study. **Your family will receive a gift card for \$25.** You may be responsible for paying state, federal, or other taxes for the payments you receive for being in this study. Taxes are not withheld from your payments.

#### What other options do I have?

If you don't want to be a part of this study, you have some other choices. You could:

 Get treatment without being in a study. You can continue to participate in EMPOWER as much or as little as you like whether or not you choose to continue to be in the study. • Take part in another study.

## How do you protect my information?

We will keep information we collect about you confidential. We will share it with others if you agree to it or when we have to do it because U.S. or State law requires it. For example, we will tell somebody if you we learn that you are hurting a child or an older person.

All information you share will be kept on a password-protected computer. We will not store your answers with your name, but instead will use an identification number.

When we publish the results of the research or talk about it in conferences, we will not use your name. If we want to use your name, we would ask you for your permission.

We may also share information about you with other researchers for future research but we will not use your name or other identifiers. We will not ask you for any additional permission.

#### Do I have to be in this study?

No, being in this study is up to you. You can say no now if you already know that you do not want to join the study. You can say yes now and if you change your mind later, you can leave the study at any time. Just tell the study staff that you no longer want to be part of it. The researchers may still use the information they had already collected about you before you withdrew from the study.

There will be no negative consequences regardless of what you decide to do. Your decision will not change the care you receive or benefits that you would normally get.

The researchers may withdraw you from participating in the research if necessary. If you or your family no longer want to participate, you may stop at any time.

#### What if I have questions?

Please feel free to ask us about anything you don't understand.

If you have questions later or if you have a problem with the study, you can call the doctor in charge of the study at **860-930-1702**.

If you have questions about your rights as a research participant, or you have complaints about this research, you call the Yale Institutional Review Boards at (203) 785-4688 or email <a href="mailto:hrpp@yale.edu">hrpp@yale.edu</a>.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time

#### **Authorization and Permission**

Your agreement, which we will document with your permission now, indicates that you heard and understand this consent form and the information presented and that you agree to be in this study.

We will provide you a copy of this assent form.

#### ENGLISH CHILD ASSENT

## <u>Child's Assent for Being in a Research Study</u> Yale-New Haven Hospital/Yale University School of Medicine

<u>Title</u>: EMPOWER Program Questions

#### Why am I here?

We are asking you to take part in a research study because we are trying to learn more about your feelings and emotions. We are inviting you to be in the study because you are participating in EMPOWER this summer.

#### Why are they doing this study?

We want to understand the EMPOWER program and how EMPOWER may change how you think about feelings and emotions.

### What will happen to me?

You will take part in a summer program by playing games, doing stretching activities, and learning about COVID-19 safety. We will also ask you questions over zoom. We'll ask the questions two different times. You may hear the same questions twice.

#### *Will the study hurt?*

You will only be participating in the program by answering questions, playing games, and doing some light stretching and breathing exercises. You will also be answering questions over zoom. There will not be anything that hurts. But if you are unsure or uncomfortable about questions or activities, you can pause or stop.

#### Will the study help me?

We hope that participating in the EMPOWER program will help your emotions and feelings, but we are not sure if it will.

#### What if I have any questions?

You can ask any questions that you have about the study. If you have a question later that you didn't think of now, you can call me at 860-930-1702 or ask me next time. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time

#### Do my parents know about this?

This study was explained to your parents and they said that you could be in it. You can talk this over with them before you decide.

#### Do I have to be in the study?

You do not have to be in the study. No one will be upset if you don't want to do this. If you don't want to be in this study, you just have to tell them. You can say yes now and change your mind later. It's up to you.

Telling us now that you are ok answering these questions on zoom (which we will write down now) means that that you agree to be in the study, and know what will happen to you. If you decide to quit the study all you have to do is tell the person in charge.

#### رضای تنامه فدی نبرای شکت اظالشان در مطلع متح وقی

#### پونهونطبه عل

عنوان مطلعه به راه ل دازی و ارزیهای ی کمبرن ام هی اگه ری سلانه ی و هی جلی به رای که و کمان م هاجر در جری ان هم هی ری که هی د ۱۹ می به د ۱۹ می خارج ای این نهی که و آموزش سلانه ی به رای م هاجری ن

م في قاصل عالى ريدرن ام ه ش خصى كه ههى ي ولا ي نت في ق ست (: جواعا روزندر ك، MD MHS

(333 Cedar St. New Haven, CT)

شمارهماس: 8609301702

#### خلاصده مطلع متقع عقاتى:

- از شما وفرزنتان مخوای کم به طینبرن ام متر و وی د.
- ددف از نان مطلع مت تحققهای ارزیهای برنام ه ای استک ه خلو اده شما در آن اش راک خوا ف د داست ببرنام ه مگوینام EMPOWER مهاد و ارزیهای آنها ازبرنام ه در جری ازبرنام ه و بعد ازبرنام ه ال جام ههاد .
- دون ظرس نجی از طری ق زوم همر اب ش ارک ت درب رن ام متعلی کی مشم اری از داری د ( لازم س تب ات وجه و متص میم خود میتورای میتون در ای در ای میتون می در ای میتون می در ای میتون در ای در ای میتون در ای در ای میتون در ای در ای در ای میتون در ای در ای میتون در ای
  - تلت دربرنام هنیزب شی از عن مطلع ه است.
- سروی وببررسی ها از طریق زومتق هیا کس اعت را دربر خوا هنگ فی تبتم هن ات عارب برنام ه هر ففت ه شامل سهبار هدن رودر رو و یک میار هم از طریق زوم طی دو ففت ه ل جام خوا ف دشد.

برای افزیرک در بین مطلع ه خطرات هم وجود دارد. خطرات شامل پلی شه های محنوری دفی طویت های شخص ی یا دوستن نافی تون های محنوری و این از برخی از فسطی ته او و النامی که پرسی ده خوا ف د شد.

عان مطلعه م کنکه ها جرفت عیب رایف رزندشمان نایت مبلاد اما عان مطلعه م کنبه کسرایک مبرنامه های نفریاه و را دربخشه تول فیدسازی دربان می دربان می دربان دربان دربان می دربان دربان می دربان دربا

گنون ه های هگری روزبر ای فرزندشما و جود دارن که خارج از طرنت بی هی شرند. لازمی روستک فرزندشما در طرنت بی قر اککند د خاگر شرم دربرن ام متول فردس از ی شرکت کونید.

### چرااینت قیق مطلعتیبراف رزند من وشکش میشود؟

از آن جازی فرزندشماق الا دربرنام متول نه سازی نابتر اکنموده ما ازفرزندشما می خوای یک در باین برنام متخصی مطل علی به نرش کست نظید. در مطلع متخصصت می از باین برنام مبشن د. در مطلع متخصصت می شاکست و دربرنام ه ارزی بای تول و بستان می از باین برنام مبشن د. در مطلع متخصصت می از باین برنام مبشن د. در مطلع متخصصت می از باین برنام مبشن د. در مطلع متخصصت می از باین برنام مبشن د. در مطلع می از باین برنام می نود دربرنام می نود دربرنام می نود دربرنام از باین برنام می نود دربرنام در باین برنام می نود دربرنام می نود دربرنام در باین برنام می نود دربرنام در باین برنام در باین برنام می نود دربرنام در باین برنام می نود دربرنام در باین برنام می نود در باین برنام می نود دربرنام می نود در باین برنام می نود در برنام می نود در باین برنام می نود در برنام می نود در برنام می نود در برنام می نود در برنام می نود برنام می نود در برنام می نود در برنام می نود برنام می نود در برنام می نود برنام برنام می نود برنام می نود برنام می نود برنام می نود برنام می نود برنام می نود برنام می نود برنام برنا

## چ کسی مصرفای نت فی ق راپرداخت میکند؟

ى كادرى كالمادمى كالماران اخال، الهرتينى و تاملى صرحت/ مركز ملى يهيش فت علومكا لوردى (NIH/NCATS)، وپ و فتوزيهال عارفت بخى ق را مركون د. تام الماران اخال، الهرتين و مناور بهال عارفت بخى ق را

#### چ کسرانی بی گری ای نت ای ق را حلی سم ی نند؟

الناز الهت از طرنت في حجات ميكند.

## این مطلعه دربارهچیست؟

هدف این مطلعه ارزیبیای و اجرایب رنامه ملستکه خلواده شما در آن نامیت راک خوا هدن مود وی ا همها نامیت اکن موده ان که معروفیه معروفیه معروفیه معروفیه به برنام متول بید سازی EMPOWER میمیش د.

#### فنورزند منمی خوه ی د چ کاری ان جام د هد و چه مدتای نیارن امه طول می کشد؟

گسرشمب کودکت ان اجاز مبدی ستا در طرزب رن ام شهر اککن د، طرز فای افتای ستک مپیش می غَد: ما از آن ها از طوی ق زوم واله ی را می پرسی که هر شها می برسی که فران برسی که و اله ی در مجموع دوس اعتشما و پرسی که هر می کوش مطرز کواه می برن می دوس اعتشما و کوک ان شما را خوا هنگ فرت برن به فرف می برن ام ه ای برن که می مدت سه ساعته و شکل می وری و به مدت ۱ ساعت ه رفته از طوی و دو مدر طول دو فقه میگز از خوا هدشد.

#### ریس ک دا وراد حتی داینشی ازای نهرنام مبرایشلتر اکسننگان چیست؟

## من چگون ه خوا ه متوانس تدر موردریس ک ه ای تازه و مغیومات م ه مای نت ای قادی خص که نم؟

گسکدام چلومات جهد راجعبه لین تخوق بسته ی آوری که مکن استن ظرش ما را در ریاط مبا اثبتر اکک و دکشما در لی زب برن ام متغیر بده د، ماشما را در جری ان خوای مگذشت.

#### چون داین تهیق می توان ب کودک من فمی بسد ؟

ب آمویخان در موردص حت وسلامتهای از طری قیب رزامه EMPOWER کو دکشما مکه ن ملت فی دمبرس د وی ا مهن رس د.

### چطوراین ته قی قب مسرای ر مردخلی دهمی رسراند؟

فعلده ایکه از عاربت خی قبه دلش و مردم می رسد، یک گما ه یه بعقری راج عب ف وعل برنام ه EMPOWER و تلیت راک عارب برنام هبا هگر ان بست ما خوا هد داد.

## برایشلتراککردن درای نبرنامه فی کدام فن میاختهشود؟

شملبرای نامیتر اکفرزن ستان در علیبرن ام ه مهورب مهرداخت می چه هنین ه ایری می بین دین ها مهرف می قید مهر ف می رف ت می مک امهوت رک ه از طری ق زوم ب خاطر را جام مهراهی ه های برن ام ه EMPOWER لازم تهیشد، خوا ه به ود.

## ق ابرای کودک احکدام معشی بلبتشل تراکشان درای نیرن ام میرداخت خوا ددشد؟

کودکشما هیچولی رابطبت شیتر اکشان در عانهبرنامه درهاستنخوا فیکرد اماشملطبت حضور در هرسرویکه از طویق زوم ال جام هیاهبه ارزش 25 اللرگفیمتکارت درهاست خواهیکرد.

## اگت صعی کیس ری مک مب حد د اجازه شکت درای نیس رنامه ران هیم، چ گون ه های را در اینی از خواهی مدشت؟

به جای التراکنمودن در طرنت خی قشما فگرگ زین ه ها مه داود.

#### كودكشما عنونكه:

- دربرنامه EMPOWERش کتکن شبدون وانکه درت وی قس مجگیرد.
  - دې چې ق مگری شرکت ن چاد.

## چطورشما می وماتک ودک ام را امن و محرمنگ دداری مین ید؟

تمام علی مانتکه درب ارف رزندشما جمع آوری میشود ار طرف مه طور محرم نگه داری بهشود. طبق قولی ن آمریک این المبار و است ما علی و مانتف رزنت از با در خولس تکنی دبه طور شال مکسی را در جری ان می مرفیم گلر بان شری ک میشود وی ا مه در صوری که قران علی ته حده و دولت از ما در خولس تکنی دبه طور شال مکسی را در جری ان می مرفیم گلریف میمک کسی به افظلی ها بازرگلی ال کن شرر میرس ان در جری ان می مرفیم گلریف میمک کسی به افظلی ها بازرگلی ال کن شرر میرس ان در جری ان می مرفیم گلریف میمک کسی به افظلی می بازرگلی ال کن شرور میرس ان در خواند کنید به میمک کسی به افظلی می بازرگلی ال کنی در میرس ان در خوان می در می میشود کنید به می می بازرگلی ال کنی در می در می در می در کنید به می در می در می در کنید به می در می در کنید به می در می در می در کنید به می در می در می در کنید به می در می در می در کنید به می در می در کنید به می در می در می در کنید به می در می در کنید به می در کنید به می در می در کنید به می در کنید به می در می در کنید به می در کنید به می در می در کنید به می در کنید به می در کنید به می در می در کنید به می در کنید به می در کنید به در می در کنید به میگذارد به می در می در کنید به می در کنید به می در کنید به می در کنید به می در کنید به در کنید به در کنید به در کنید به در کنید به می در کنید به می در کنید به در کنید

عربت تی قب سرطی کی و اور مل و از مؤرس مهلیب ویش داده شده است. م تی ن دارای عارک و اوی ن میتوران د اطلاعات، الرن ادی ا ن مون و وای دادرس عف در ال و الله علی می در ال دادرس عف در ال و الله علی می کفوری، اداری قرار و نگذاری می در ا

گواهی محرمل هبودن برای جل گیری از فلش ای آن مواردی که قرار و نفیدر ال، طالت ی در موردس و علیق اده و فغلت از کودکی الم بریب رس ال در نبه خودی افک ران ال زامی م که نید، ملیق ادهن خوا مدشد.

## كدام اطلاعتى را در موريكودك ام در لىن مطلعه جمع آورى خوا فيكرد؟

در مورد قرانون حریم ضروصی و خیروق شخصی شما میتولی ب هاس رحریم ضروصی میل در 5919-432-203 صیحت کیلید. علی و مات شخصی رک م ما درب ار فرزن د شما و لل ت صحی شان جمع آوری مین هام و از آن ملیق اده مین هام شام ل:

- تحقیقات مطل علی میشده بدون کرن ام و شامل جوبانته و االت سروی هیشد. این و الت سروی شامل و االت دربار فشار روح کفیت زنگی فیتار های صحی و ف ممشان از کید ۱۹ هیشد.
  - لرن ادیکه در جری ارن چیق از طری قیت ماس فین ویت می مشده راد.
  - المرن ادی راجع، مضری کودکشم ا دربرن امه EMPOWER

#### شما چون ه از اطلاعات و دک منسل شاده وبا ی گراش ری کم هرازی د؟

مطلقیتشری حالتک و در بیان رضرهات نام و مطلع کر فید ما علی و مانت رزند شما را ملیهاده خوای مکرد.

## شهد مم عل وماتف رزندشما رابا:

- هارت ف صحت و خدماته شری کسازی م.
- بان چلن دهپو فتو ری لهبابرن ام ه فحاظت مطلع التعبشری ی ل وبابور هبرسی ساز ملی وباک چه مبرس یک ه رایس ان ۱۰ در آن مطلع ات شهر ند.
   شهر اک کهی رن د و بی ن مطلع ات از طرف هبور همی ق و مرقب ترفی ترفی ند.
  - باک ایکن ازبخش صحیکه خدمات صحی رابر ایف رزندشما میرس ایند و در عان مطاعه ارتب اط دارند.
    - با مخفق نطن لى عان مطلع ها مخفق نه محار وسهار مخفق ن مهوطه.
      - با هما فی کوننده و الجن ایه تیم مطل الله

با ه کار انبخش اطلاعات و اهنای ارقام وبور د مرقبتای و نظیر قهامات با اسلاح تکه از تطبی قبرن ام ه مرقبت میکند.
 مان طابت تالاش خود را میکنی کشما را اطهن انب دی یک ه خل و ماتف رزن دشما خصوص یبقای خوا فاد مل د اما گلر ما چل و ماتف رزن دشما را همرای کسر شیکه قال و ن حریم شخصی را فهال نویکون د در آن فیگام چل و ماتف رزن دشما فیگرت و با فیل و ن فیظ حریم شخصی م خلطت نخوا فادشد. ل فیل و ماتف رزن دشم ابنقار و افت رزیگ مداری شرو د با و می داری شرو د او می داری شرو د با و بازی ای می داری شرو د از طان ها موفق تن ام و می د فیک متم ام علی و ماتف رزن دشم ا را م حرم نگ مداری میکن ند.

## چراللی د منبرای میلولهتی که درای نسن د در جشده است، موفلق تن ایم ؟

با موفاق تعان سن دشم ابر ای بی متحقق بای اجازه می دی یک م علی و مهای شرح داده شده را در علی مطلع ه ملوق ساده ن طهان شون که علی و مهای شروی و ماسکه مرتب طب و این در می تعرب و این در می توسی و می از دارن در در می از در در می می می در می می می می می می می در اداری د.

علی و مات صرح ف رزن مت از که در جدوری و عیش ان عهد در اداری د.

## اگفکر من در موردای نهرن ام مغیرکرد چی؟

صلاحی ت طف ده و شری کس ایجن علی و مات صرح ف رزندشم که در جری ان شتر اک غش ان درب رنام ه جمع آوری شده می چگاه ی قضی نوش و د. در چند شما میت وافی در از من ام خود را در زمل ی پس بگی بی دب رای پس گفت نوش در من با جازه ن ام همرای کس و خود را در زمل ی پس بگی بی دب رای پس گفت نوش در من با جازه ن ام در ای در من با می انش تن رشت و ب و با در سیف برستی د:

Julia Rosenberg, 333 Cedar Street, New Haven the Yale University, New Haven, CT 06520

## چی خوا ددش داگر من خول ت مبش که تین اعن لهیم وی اب مثل تر اکف در زندهی با ازت مامش در نهر نام ه جتم مبد مم؟

طین کا در صلاحی تشما مل ستک می فیرین تنان اجاز میدی که دربین امه تایی را که کند. شما حق فین خاب را داری که اجاز میدی دی اجازه ندی د. شما میتورای فی کند از میترسی و به خدمات صرف در این میترسی و میگر میترب دی د. می و میگر مین می می در از میتن خوا مد.

ازفر زندشما خوبلت ه خوا هدشدک ه رض بیتن ام ه راسی ای مکن ستا در عی نهبرن ام ه شامل شود. گدوفر زن ستان نخوا هد در عی نببرن ام ه شور اکن جلد آن ها در عی نببرن ام ها و جود رض بیتشما هم شبت و راجیترن خوا ف دشد. دلی ل عانکه چرفر زن ستان کی خوا هد در عی نببرن ام هش کستکن د از شما پرسی ده ن خوا ه دشد.

با لمان و جود هم مفر زندشما رابه طور لمویندار در مان خوای کسر وی ا هجه در خواست شمله که ای کی مهدوطه وی ا هم نکستار ناش ان مراب امراب می میدان می مهدون در رابط فر زندشما همراب امراب می میدان و می میدان در رابط فر زندشما همراب اکستار ناش ان وی ا هم المین در دادن خوا هد مشرت.

برای خار جشدن از طرنبرنامه ههورای د وگاه خواس مبلای دا ایخن ای طرنبرنامه مطلع مت هی درتماس شهد م الاگورزندان شخص بسازدی و درای نورند و درای نورن ام شلتر اکسند.

## با مغیومات جمع آوری شده دربارفسرزن من چی خوا هدش داگرایش انب شل تر اک خود درای نهرن ام متوف فبده ند؟

فرزندشما مهاور شهر اک خود دربرنام متول فیدسازی ادام مبد مدگرچ مشملخوا میدکه دربرنامه والت از طری ق زوم خانم مبدهد. شما مهاور همتول سای دریفات چلو ماتفرزن متان رابعد از آلکه جمع آوری گری ن در لبکید.

#### اگرسولی فلت مبلی بلی بب متماسشوم؟

شما عهاواليد آزادل و درباره ورجهز يك ون مدالي دسوالكرفيد.

گر الج بل أشم كدامسولاى نتات مبترى دى ك مبار مطلاع مت تحقق بلى نتائج مبترى د مهتورلى د م قرق طل لى يبرن ام م م عن شمار و زنگ مبزى د م

گىر درباره خىوقفىرزنىتانىبە مىڭ ئىتىرككىنىدە در يانبىرنام كىداس، والى دئىت مىئىرىدى يايىكە دربار مەخچىق دئىت مىئىرىد مەولىد ب مبور دىبرسى يەتچىقىلەر يىلى يارىكىلىدىنىد 203-785-4688 Email: hrpp@yale.edu.

#### ل<u>تی ی دی و اجازه</u>

مولق تشف اهی شم اهی نکان ون در جس نو دال ال تعبر آن هی ن که ن که ن که مشامل می این می و شد ای د و ب ف رزند تان اجازه دای که مشامل علی با نام هم مطل علی تا که مطل علی تا نام د می تا نام د مطل علی تا نام د می تا نام د ت

برایشمای کیپای بینسند راتی ه خوای کرد.

#### DARI ADOLESCENT ASSENT

# توفقن لم م بن کس الان مبنى برشل تراک و ی ک مطلع م تقع عقالت ی ک مطلع م تقع عقالت ی ک مطلع م تقع عقالت کا در ا

**عنوانتی ی ق:** اجرا و ارزهیای کسبرن امه آموزش احتماعی- هرجای و سلامتی برط کودک از پینا فده در جری ان مه گیری کو هید- ۱۹: Empower برن امه هیجان مای خارج ای اعینی ک و هید- ۱۹: Empower برن امه هیجان مای خارج ای اعینی ک و هید- ۱۹:

شماره تماس: 1702-930

## چرا مراين جا ام؟

- ما ازش ما می خوای ها دری ک مطل عت خوقهای شن رک کنی د.
- عارن جی قی قی جرب مشما را دربرن ام متبلست ان بررس ع خولد کرد.
- طین لچس منق رهای کس اعت رقت را در دو مرق عیت جده بله درب رمیگی رد، ممرامباس و الای یک از طری ق زوم پرسی ده می شود.
  - طین جلس هبه م چی شنب راکشم ا دربرن ام متبلست الی EMPOWER بلیت که شامل فعته ی ۳س اعت جلس ه خضوری و ۱س اعت جلس ه از طری ق زوم برای مدت دو فعته میبش د.
    - ى ل فورم الوقون امه، مطلعه عق تحقیلی را وس مهشم ارا در آن وضوی ح می د مد.
    - لفاب، قىتىب خورلىد. مر الدازه قتى رك مضرورت دارىد، مى توراتى د المقاه كى د.
    - له ازكار في دان ت في در مورد مر آن چه راجعبه عان ت في قنمي دالي د سول كنهد.
      - شما مه تورفید مهن االی ا مر زمانی در جری انت تی قسوال مطرح کرید.
        - گار درت قهق شهراک مم میکنهد، میه ولی سبحداً مهر فشهد.
          - شما هر زرهای که خوالرن مبشری د میتورای متخصق رات کوفی د
    - مابهپدر و مادرشما مم در خوبلست خولج کرستاشما رابه شهراک در بین تهیق اجازه د فد.

## چرالىن تىقىق بلى من يۇن دادشدە ست؟

ازش ما می خوا میمتا در بین مطلاعت خوقهای س مهبگی رید نی را قرار بل ست**شما وفلم ول شما و ی کسون لم متامی سانی** ش**رات راکک ری د.** 

ما در جهتجه کودکه ای استی که در بی نبون ام ه شرق اکسرده از در حدود مجموعاً ۷۰ فرت در بی نوت کی قس مم کسی رن د و بیشت ربی آموزن دکه بی نور نام مبر ای شما و ف ای لشما کی ون نور سرت .

## تخىق در مورد چە الست؟

هدف ت خیق این الدیت کمبرنامه ی رکمه قرار الدی تفلم الدین شما در آنشل تراکسنندو ی اشت راکمکرده ارفکه بنام بون امه EMPOWER و بشد، را از اب کیند.

## در ج طن تخییق چانفیق بیش خوا دد آمد؟

اگرش ما موفلق بشی ها در طین تخیق شن رک کونید، طین فلقیلی لات کمپیش خوا دد آمد شم به والاتی در ج مانی دو مصلح به مصلح به جنگان از طوی ق زوم، جواب خوله ی داد. مااز شما در مورد احس اس و می جن اسس وال خوله ی مکرد. شما در یک بون له د تلمین تان مشل تراک خوله ی در که بازی کردن کم می پروژه های رس امی، آموزش راج به صرحت سال مسی، نک ات منطقت یک وی د ۱۹ وی جن اسش امل آن بون امه لات.

## من برای چه مدت دارین تخییق ی بشم؟

شما ۲ لجسه از طریق زوم خواه د نشبتکه هرکدام آنهتق هائی کساعت را دربسر خوا هنگ فیت بی نبه اضاف مبرن امه ای لمرت کسه مدت ۱ساعت هر فعته از طریق زوم در طول چهار فعته مدت ۱ساعت هر فعته از طریق زوم در طول چهار فعته گذار خوا هدشد.

## خطراتاحتملفين تتحق چيست؟

## چگون من من ومات جيد و مهم راج باهن تتحيق البست بي آورم؟

اگرما ک دام چل و مات جی د راجعبه طریق تجی قب بسته بی آوی مک مکن استن ظرش ما را در رباط مبا المت راک در طریب رن امه ت غیرب ده د، ماشما و و ال مینشما را در جری ان خوا می گذارت.

## چگون ه چ توانای تقیق به من ی کسان ی ی گرفمی تمامشود؟

## آی الل تراک دری ن تحیق زهین های برای من خوا هد داست؟

شماضرورتنداه هابرای شهراک در طرف خیق قبولبدی دبتن ها هنون ها کمبرای شما وجود دارد هنون فت و آمد شما خوا هبود.

## آی او صور تشل تراک داری بون له برای من معاش خواهن دیرداخت؟

شما در صورت شهر اک در عارب برنامه م عاشن خوا ی د دشت **فلمی ل شم ی که ای تخه ۲۵ دلی بست خواهن آورد.** شما مهره وله پر داختم الهات وله ی فلتی ف درالی و هگرم الهات که رویه پوله ست آورده از عارب برنامه وضع می شود، خوای د بود. مالی ه ازبوله پر داخت میشم از قبالت ای هنمی شود.

## منی یکر چ مکینه دا داختی ار دارم؟

اگرشمانمی خواهی در بی ن تخیق شهرک کره بستی ی گنون ه های هگر مم در ایخی ارشما است. شرما میتورهی د:

- بدون شنراک درت خیق مه حت داوی قر اربگی ید. شم ای تان ی بشل ترک تان در EMPOWERبه
   صورتکم ی تری اد، هگون که خود شم ا دوس باشی ته بشل ی د، ادامه هی د، گلو ب شل تراک داری ن تقحی ق ادامه به ی ی خیر.
  - دربرنامه هگری شترک کیفد.

## شم چگونه از من ومات من مخلطت محانید؟

عل و مهتی که از شرما جمع آوی می کنهم را محرم نگ هیدای م. در صورتی آن عل و مات رابا هگرانش ی ک خولی م کرد که شرم الموفقت دارت می از هم ما مهور ربشی مک قراشی که بسان مبخ اطریک قران و نالات ست دری افرات بخی ن در خوالیت در صورتی که میدای مشرد به طور مثال مما کسی را در جری ان خواهی گذشت در صورتی که بدای مشرم به کودکی ای ک سرالی خواهی گذشت در می رس الی د. سرالی خد می در می رس الی د.

ت مام چل و تملی ک مش ماب ماش ری ک می سازی د دری ک که بچی و تری ک میسور د داشت مبش درگ مداری خوا مدش د. ما جواب های شرم ا و با اذک رن امش ما ذخی روزم می کونی مبالک هازی کش ماره نش خصر کونن دمبر رای ذخی روزم می کونی مبالک هازی کش ماره نش خصر کونن دمبر رای ذخی روزم می کونی مبالک هازی کشرد.

ز مرایک موزی جمت بخی ق رازش رمی کنهم وی ا درکی رابس ی راج عبه آن حرف می زریم، ن امش ما را ذک ن می کنهم اگرب خوای م ن امش ما ریاه کاربب کی از شم ا اجازه خولیم گفت.

مهن لمرت چلوماتشما رابرای تخصی قرآن ده با هگر مخقهن شری کسازی م گرن امشما و هگر ش خسالت تان را لمیقاده ن خوط م کرد. از شرما اجاز ضل اف ی در خولم بتن می کنهم.

## عَى ا من من من من المن در لىنت على النيت الكنام؟

هریتص هم میک هشم المگی هی د هی چک داهی امد فه می نخوا هد دلاست بتص هم هشم ا روی ت و جه و انتی ازبلی ک هشم ا معمو لأب ست می آو ها متنقی ری نخوا هد دلاست.

م ق ق مكن در صورت ضرورت شما را ازت قى قبىر ف كند. كلر شلمى فلمى تاوى كى نخولى كدر تولى كالمن كا

## گرسول وشاته بشم چکانم؟

لظاً در مورد در چیزیک منمی دراید آزادل ه از ملبپرسید.

گرشملىعداً سولاى مى دائت مىشىدى الاركىلى يەك تورى دائت مىشىد، مىتورلىد، مىتورلىد، مىتورلىدى مىدۇلت تىق قىلىمار دە 1702-گىرشمار دە 1702-860-مىماسىشى د.

اگرشما فی چیشی ک البتالک کون ده تخیق در مورد خی و قیتان سوالی داری مورد، وی اشکای در رباطمبه علی نیت خیق داریت بازی د بابور هبررسی البیت ی و تخیل باشماره 4668-203(به تماسشی د هی ابه عیم ل آدر س hrpp@yale.edu عیم ل ارسول کید. 

## لم<u>قى ى دى</u> و اجازه

موفلق تـشما ركـمبا اجازهشما مهـعلاً مهتن د محكولهم، رشان مى د ەك مشما لىرىف و رهتوفلقىن امه و مافيومات ارىئ مشده را شرىھ دو ف مىھدە كىد و شرما موفلىق لمەتكەت درىل رىت تىچى قابىشى د.

ملبهشم له کدلهی ل فورم الفقن امه راتیمه می کریم.

#### DARI CHILD ASSENT

# توفقین ا محویک مبنی برشل تراک در مطلع ه تخ وقاتی شفاخ نی ی ل نوو واین/ پونتون طی ی ی ل

## عى وان: سول هاى برنامه Empower

## من چراطن جا ام؟

از شما خوا هان المیتی بتا دری ک مطلع می تحققی شرکت نظی د. چون می خوا می بتا در مورد احمی اسات و می جان های شما چل و ما تعبی بت به تعدید کرد. EMPOWER شورک کرد.

## چرا آن ها لینت خص را ال جام می د فد؟

ما می خواهیم در مور بسبرن امه EMPOWER و تانک، مجلون، EMPOWER طرزف کسرش ما رازیس سب الحرماس ات و می جل انت خی رخوا دد داد کم گا می پی لاکنهی م

## قرار س جفاق عبرای منهیش ود؟

شما دری کمبرنام متبلسته ای شهراک خولی کسرد کسمبانی کسردن، اجرای حرکست کششی و علی و مات راج عب منکات مغلقتنی کسوهید-۱۹شامل به نیب بن امل ملت. ما از شماس وال های را از طری ق زوم خوای مهرسی دبس االت دوب ار در دو زمان منخلف از شمه پرسی ده خوا مدشد شما آن س االت را دوب ار خوای دشرهی د.

#### قى الى نت عقى كدامض ررى خوا مد دارت؟

شما در طین برن ام مبعب عضی س ال تعبیل خواهی د داد بازی خوط هد کرد، کهوات کشش ی و تف س آزاد را اجرا خواهی د کرد شما مریخ ان بعب عضی س اللت از طری ق زو مهیل خواهی د دادبیس ک دام موض و عین خوا معبو ستاب مشما ضرر برس ال کرشم الله گراگ در مورد س وال مو فعالی ت ه ام طوئ وی اراحتری بی بی در می توانی که ادام من دی وی اتوق کونی د.

## غياط نه تهي قهاراي منكك مي كند؟

ای د داری مت المت و این درب رن ام EMPOWERبه می جل ات و احس استشمال کو کند، اما مطعی ن نی میک می بی ن خوا مد شرد

#### اگر سرو الى دىلرت مېلاس جمهاد كن م؟

شما مهتورهی دگدر سولای در موره تحقیق دافت مبشی هبپرسی د. گدرب رای شمابعداً سولای پی داشت فع الله و نه من شمان هرسد مهتورهی در موره تحقیق دافت مبشی هبپرسی د. گدرب رای شماب عداست و میتورهی در می الزرج می التانی به سرمان و التان می الزرج می التانی می التانی می التان می التان می در هبر می التان و بستان و این و بستان و بست

#### غياو الهن من در عين مورد مي دراند؟

علىنت تى قب دو الى ن شمك وضرى حداده شده و راها گفته لادكه مى تورانى در آن الت راك كى دار شما مى توراد قبال از بان ك م كان كى در قان مورد با قريبا قريبا قريبا كى دى در يان مورد با قريبا قريبا كى دى دى يان مورد با قريبا قريبا قريبا كى دى دى يان مورد با قريبا

#### في ا من بعلد در علي المنت و المناسم؟

شُم اُ مهتولید که در این تخصی قس مهنگههد. کسی نار احتن خوا مدشداگ رشما اثنیتر اک نکیلی د اگر شمان می خولیع که در این تخصی قب اثری دصر فسیه آن ملگهها د. مهتولی فسعالاً ای یه گهری د وبعداًن ظرت ان رات نجی ر دی دب ه خودشمات فی قدار د. طن که ملب هس وال های ما در زوم جواب می دی دب بده طین م قهی لمریت که شما موفساق لموتید که در مطل عجماق ی ب مرای دائی که قرار لمرت چمپی شره بویلی د اگر شر ماتص هم بگیری د که ترخی قرات رک کونی د سیمام مجیزی که بطی بدیلی د طین لمریت که به شخص مری و لوبگ هی د

## د و څوړنی د مطلع اپ اره د ولاینو اجازه و لقی یدی

#### د ول طبى ونتون

د **مطلعی عنوان:** د CoVID-9آپر اخ مرضوپر مالی د کهوال و مشوطه لپاره د هور<u>یمان</u>ې اوټولهیز - احرماریشي زه کړې برنامچل*يي ک*ول او ارزونه: Empower

)د مه اجرون لپاره کاون ک اوسال منعلی م خ خوب د اص الدیدوبرن امه (

اصلي څون ویه ) د څوک چې دې څوړنې مراوی تاري (: چای اروزن رک MD MHS

(333 Cedar St, New Haven, CT)

د تهاون شوی ده: 860-930-1702

## د څوړني مطلع خالصه:

- مون ریت الس و او سیت الس و مل و می و خود اینه کو و چی مون ریس ره د دې څین دویطه اله عه کې کیدو زوکېړی.
- د دې څه رړندوی، مطاعی هدف د ه غې ځېروڼې ار زویلیی ده چېسټلو کورڼیکی، کېډن کوی، او ویاې کېړی و ي،
   ار زویلی یم ځې کېپه جرویل کې او وروټه د ګېډون څخه اخولی کېږي.
- دوېسروې)نظر وکول (د زو له الريپدې او چې کېښروري دي. )ټر څوبې له پځلېپ وکېړې د مطاعي ته دوام وکېړي.
  - کدن کولپدیپوکارم کی بخاله د مطاعی موبخش دی.
  - داسرویبه دو هسای لپاره ویپه درېځلي خسوري، او اللان د زو له الرې دوځلې په دوه فمن کې د
- ګډونېه دېمطالعه کيوب ځښې خطرات لري. دا خطرات بېځښورنگونوي اچالشون څخهبر خمن يي لکه په چښوري خپرون کي چښوري خپرون کي چښورل، اوي ا بېځښېسوالون د مطرح کي دو څخه ناراخي.
- دا مطل عمبر على عسلس و مثري م ك و مفعل ده رؤلرى. او ببر على د ه غوكس رأو لهار ه فهي ده و وسي چى د Empower په شان مربه به يوگ را ده و علاق من ه وي.
- د دې څېړنې نهب فغېرستملس و څښوم از نوربل لټخاب م کولی شی ستملس و مځل و مېطاده ن ده چې دی څخه و کې کېډون
   وکېږي که مېملل و د Empower غېږد ی ځېړنو کې ګډن کېوي کې دی.
- خانته او خیال مشومتمپدې خوښوکی ګډن کولسټلسو بنځله خوښه دهبتللو کویشۍ چی خوښې کړی دې
   پاره اجازه وکړی او ریوڼه کړی. او هکله ځیا فکرتنبهدلون وکویشی. هر اټخاب مو چېوکړ،سټلسو مشومېه خیالصحی مراق له السه و رزکړي ان ه کومېلولونی حق او فهاد.

## ولى دا مطلعه زما مش و سه و ران د كى ي ي ؟

مهن برسټنلسو د مېشوم څخه غواړو چېپه دې څړېنه کسميسرخه ولځلي ځکه چېسټنلسو مېشوم د Empowerپوګیلم کسی ګیډن کسو ي. مهن بر د ۳ ګیمورځیو او ۷۵ مېشو مړلوپ های کسیمیوت ر څو د دې څړېن یېسر خه شیمیپ دیمپ پګیلم کسیډ ګیډون څخه مځ یی او وروسټه هېوګام څخه اړیملي کولوپ هشمول.

## څوک د زکړ ښيارپ سی و کو ي؟

د اکادی کسی هیئری کستوانی ه، دصحت ملی اندینی و به کاربر دی سرفان س مپر منح ک ملی مرکز (NIH/NCATS) او دی ل پ و قتون دی تحق فی ایار میکن و کوی ؟

## څوک د دی مطلع اي نو مال يې چمتوکوي؟

الهن از لاي د دې مطاعي لپاره مات چې کوي.

## مطلعه د څهشي په مکله ده؟

دې مطاعې دف هبرنامې لي کول او ار زون ده چې تالو کورنۍ بکېې کډن کو يې اې کېړۍ دی، چې د Empower په نو هيې ژندل شو ي ده.

## تىلى و زما د مىشوم څخە څەوغىتىن كوى او څومرە ىخت بونىسى؟

## د برخ ه ځیتنی خطرون ه و نالحتونیک و می دی؟

كىمتىلىرو او كىاستىلىرو مېلىرومازىپ يېچېد وكىدى ئې چېپىدې مطالع، كىمبېىر خە ولځلىي ئىتىلىرو او كىاستېلىرو مېلىرومان مېكىن د رزېچ يېنوسىرە مخشىمىپ شىمىخىي فىعالىقتىرىق كىمبېىر خە المچىيىتىلىق كېمشىمىخىي فىعالىقتىرىق كىمېن، ئو كىما ئىپسىنتىلىشىوي ئىمنى يېپىنىتىنو څخەن اراقتىي.

د محري له السه وركولو الحامال خطرشتون لري.

## <u>ه زیه څنګ د نوي خطونۍ یا د مطلع په اړه م همو مځې ولمت په اړ و پوه ی وم؟</u>

مو رب متلال وت و ويلي که چهرې موريک و مڼو ي ځلومات زه کېړوچې کولۍ شي ستلال و مثل و مپه دې څه يڼه ک بېبر خه اخهتال وي. اخهتال وي. اخهتال وي. د د زيالي کېړي.

## مطعه خنگه ممكن زما مشوهبته ورسوي؟

ستملس و مشرو شری فی فی ده و محلی می اولی به نظامی و مطاعی شخه، د رو نځی او هور وانی او د کول ل ه ال رې د Empower د پوه کار ام څخه.

## <u>څنګه مطلعمممکن نورو څکو تګټه ورسوي؟</u>

سُرطنس اونوروخلکونه کېدایشي دښمپو هاويشامل وي چې د EMPOWERبورامې ګټې او او څځکه دلبرنامه نوروسرهشوکمول الرې.

## 

تىلىرو اېزىرلىلىرى خېل مائىرو مېمىدى څېېنە كىمبىر خە الخىيىتى لېارە لەبست وكېړى.ىوازې لەبست مېرالىمپورت او د EMPOWERبرنامېتە د رىكك او د زوم كموي كىمشامل دي.

## ای ازما مشوم نګډول پاره معاش و کولی ی دی؟

ستخلسو مېشومت مبويدې څخېړه کــې هــبـرخې المجيښتي لېـار مېيسېنه وکـــلي کــيږي ، کېـرتــنلــيوبـه د زومسر يي کــــېـبـر خه المچيښتينې د هر مثملل لېـاره )د څخال مېشــومسرد( د 25ډالـروالـۍ کــارت دکـــړلـشـي.

## زمولنت خبون، څه دیکه و دیک و دیک د و دیک د و دیک او دی خون کی د و دی خون کی د و دی خون کی د و دی کاره و داد کاره و د

په دې څون کې د ګډون پرځای ماس ځونې نور له خپون لرئ.

ستساس و مانس كولىشي:

- پر ځای د مطّاعېپه Empowerي ګډن کول.
  - پیمال مطالعه کیمیسر خه اخیسال.

## تاوب، خنگ زما د مشوم مل ومات خوندی و خصوصی وراتی؟

موربب سيتلسو د مټلومپ اړه ريټول شوي عل ومات محرم وسيتو . مورببه دا دنوروسره شوکک کېړ کمتلسو موفل ق کملت ککه له چې مورببطد دلترس و کېړو ځکه چې د مټحده ا االت که االت ورته اړيا لري. د مټالپمتوګه ، مورب کې و چاته وولیو که ههرې موربپو مشو چې دو څوک مټلوم که الوی سړيټ ه که ان رسوي.

کــله چې موږ د څیړڼېپېالې خېرووييله کـفېراښون کــې د دېپه اړه و غړېږو ، موږب،سټملسو د مېلسومهنوم نوه کــار و. کــه موږ غواړو د دوینو هرکــاروو ، موږبه ل.متــلسو دواړو څخه د اجازه لی کــ غوښتونه ولځلو.

موږيب سيټلسو د ماشومپه اړه ځلومات د سالونځي څهري لپارهنورو څهړونځوسره ممشوکۍ کېړو ګهر موږيبه د هغصا هغېنومېانورشن اخت وکونځيشوان ونه کاروو. موږيه ل متلاو څه د کوملافي اجازې غوښتينه ونګړو.

## بدى مطلع كى به زما د مش و په اړ كوم مل ومات رتولكرئ؟

ه غه م غی و مات چې موږي د کارول و اوش وکمول و غوښته کوو د "م خلطت رو يخی ا علومات" ولي کېږي. د اد فدرالي و بلون ل خولجه خلت کېږي چې د خسوص ی جېم و بلون د حمل و رو لو بلون او ځوبلون ې) HIPAA (رو نځو نلی د د مال و رو لو بلون او ځوبلون ې) HIPAA (رو نځو نلی د د مال و رو نځو بلی د د مال و رو نځو بلی د د مال و د د د مال و د مال و د مال و د د د مال و د د مال و د د د مال و د د مال و د د د مال و د د د مال و د د د مال و د د د مال و د د د مال

- د څېړنې مطلع مبدون دنوم څخه ه هاره ي کوم چې د سرو ې سوالون و ته وکول وي. پدې سرو ې پوښتن کې د فش اری تش هش ، د ژنود کوهې ، رو نځی اچلن د ، او P-COVID اپو هې ه اړه پرښتنۍ شلی دی.
  - سوبلق نتافه بن يتمل بن وپه اړه د دېبرن امې و وبرخه ده.
  - ستاس و د مش و د ګډون سوبلق د Empower پمېرناه کې.

## تىلىھ بە زما د مشوم مىل وملە خنى، كاروى اوشى كىدى؟

مورب سيتملس و د مثل و م چل و مات د دې رض ات ف و وې که يې ان ش و ي مطلع يې رس و کولو لپ ار و ک ار و و

موږ مکنی کولیستبلسو د ملسوم ځلومات دغوسر مشرکک کېړو:

- دېټرده االټو د روغي آويشري خدملو څلگې )DHHS (ادارېسره.
- دعماله و قاون الميتازي ، دعمال السراي څه پرنې سيلنې بېرنامې او دن ادون ويا کتنې بېدورډ) ه غک د چې ه بشري برخ ه اخيست پرنځ و په اړه څه پرن ه ارزوي متمري وب کوي اون ظارت کوي (، کوم چې د څه پرنې اطاعت ډاد لخ کولو م و کولو د کولو د کال کول و م ات محرم وسيلي.
  - د رو خې لپلمل رڼې چې کورځي څوک چې د دې مطاعې په او سټلس و مشومته خدمات چې کوي.
    - د مطاعی طال می ان ورک می

- هېاران اونوريقوتوش کونکي.
- د مطاعېن اظم او د څې ړنې ښې غړي.
- د چلومه و و خون و و بن طارته و ردون و اونور د دې مطاعې دن طارت وک لري.

موړب ه غورس ره ه څوکړو چې ډاهت ر لام کړو چې سټمل و د مېش و مهاوم ات خصوص يو پهلې شي. کې ر ،که موږ د خلکوس ره چلومات خصوص يو پهلې شي. کې ر ،که موږ د خلکوس ره چلومات شوکه کې د محرومت قو اعت څه به بنو يې ،نوسټمل و د مېش و مها تب هنور د محرومت قو اعدوس ره خون دي پهلې را يې يې د مورت ، سټمل و د مېش و و او اي اش رکت يون يې په د د مېش و د

## ولى و بلي پدىسندكى مل ولتوسره موفلق اوسم؟

پدې او کې عال ملوسره ملوقه کول متلالوبه څهړونځوته اجازه وکړئ چې د دې څهړنې مطاعي لېار مېوتوه ذکر شو ي سټلالو د مال وم عال و مالتوکاروي اوافشري کېړي. دا د مې لېاره دي چې ډاهتر لاره کړو چې د دې څهړنېپورې اړون د عالومانتولو خواوت شټون لري څوک چې مېن ستخي ق مو خ لېاره ورته اړی اولري بتلالوت لحق لرئ چې د دوی رو خولی سوليق کې د ښل مال وم رو خولي عالومانته کا و ماري کا ورئ واکمپلېکې دی.

## که و خیل نظ بدلکیم نو خ به ی و ؟

د دهطال عې کې ښرخه انځيوټنې پېر مه السټلل و د مان و م روغي اع ل و مانو راغون و لو و اکسه مي ځل ه پای ته ون ه رسي د يې ه درصورت متلل و مکن هر و خت ښل اجاز ميې رته و ولځاي ال يې کېږئ.

بتىلىرو مېكىكىلە چې غوامې كىار فېدلەرتىپەيھىلوللوسىرى چىلى اروزىنىرىكىتىمچە، 333سى،درىستىرىپ ،نوي ھىھىن ئېدە تىھىلىچىو ھىن كىمى ،نوي ھىھىن ، 06520 CTتىمپە لھىللىوسىرە خېل اجاز مىمىرتە ولحلىئ.

که تعلل و ښچله اجازه و الحجیست ،نوسټملس و مېش و هېمپ دېټوان ښاري چېپ دې مطالع ه کې پېدې شي کېرپلملرن ه چې دوی د دوی له لکمټر څخه د دې مطاعې به روتر لاره کو چېدلورې ه ښال ري. د روغۍ لپه اړه ځېڅنو ي ځالوم انتسټملس و د مېشوم پېژنان کې له ه غوښتې و روسټن ه کېږي چې تملس اجازه ولځلۍ. ه غه ځالومات چې دم خه رياول شوي وي مېن اوس هم و کارول شي اون و روت ه شتخي ق مطاعې ټرپ اي په ورکې ل شي ټرڅو د مطاعې پېښې پې او اي امطاعې ن ظارت وقين ي کېړي.

## څوکه زه غواړم د مطلعلی د ای ته سی دو دمخد خیال ملل و کادون رنک یو یا یا ی ته ورس وم؟

ستملسو ښال مېلسومټه اجازه وکولوپدې څهېښه کې هېرخې المخميټولپارهسټملسو ښال لټخاب دی بتملی کولۍ شرئ د اجازه وکولو لټخابوکېړئ میکنلی کولۍ شرئ د اجازه ن ه وکولو لټخابوکېړئ.

موږيبه مي مهنځلل و د مال و مسره م ځي اري درم لن و کېړوي اسټلل و په غوينټن متلل کي اورنۍ کې الاکټرت و رام کې وچې کولي شي دا درم لنه و ډراهي زکېړي.

برخه المخييت لى ورورت مبرخ ه طبيت ل ب مستملس و د لکت ران و اوى ا دې ادارې سر مستملس و د مثل وم اړک ېې زي ان من زک ېړي.

د مطاعې څخه د تولو لپاره متملو کولۍ شئپه هر وخت کې د څېړنېښې غړيټه زنګ وو مئ او دویټه وولیال چې تملنونورن غواړئښتلان و مړلومېرخه ولځلي.

څهړورکئ يي مکمنسټملسو مټسومپه څهاڼه کې ل مبرخه المحيميتنې څخه و ملسيکه اړين وي لکه څېګه چېسټملسو مټسومپه ګنتوه کو ي دوینورنه غواړييبرخه ولځلي.

## زما د مشوم د مل ولتوسره به خصی دی ه چیری وی برخه اخی تل و دروی؟

سټىلى و مالىيم كولىشي د MPOWERعالىټين كىببىر خە ولجلىي څومرىيا لېږ خە چېتىلىو وغواړئ كىە دوى د زوم پېښتىن كىمببىر خە المچيىټىل ودروي. بتىلىق كولى،ش،ئ غوښتىنىوكىدىئ چې ھايا ھتىتچىق څخە ھىيټىلىشىيچىل، چى چالىوات رىلمول شىي.

## که و سنوبتنی ولرم نو و بلیدله چاس درای کون سم؟

مه بلي وکې رئ د هر هغه څوپه اړ پېوندې نوکې رئ چېتىلل و نهپو تەردئ. كەمتىلل و وروستې پوندې يې لىرى ئىما كەمتىلل و ھتچى قىپورې اړ رندىستېرىزە لىرئ ،نوبتىلس كولىي شى چېطىلىي څىړندوي ە ت پدې )88-880-1702 (ئىھرە زنگ وو ھئ.

كەتىلىرو د څېړزېبىر خە المچىيت يونځىيې متوګە د خېل مېلىروم چېرنوپ اړمپوينىتى لىرئ بى تىلىرو د دې څېړزېپ اړ مشكىت وان لىرئ بنوتىلىرو دىمىل رايوتتىتى و تىماكىتنى يېبور ډونوت وزنګىپ 602-785-4688 ( اوما د لىمل <u>Hepp@yale.edu.</u> بلدې تىماس ويمسى.

## واک او اجازه وکول

سټملره فی ظیمټرون چې موړیب *هې* او س **مړن**د کېړو دپاه ګستوه ک وي چېټملرو دا د رضر لیمټسریند اوټړدلی اوتعلرو خپال م**ن**سوم تمپدې مطالعه ک یې وي اجازه وکیوۍ

مو رب متسل وت د دېس ندی و کمپلي د کړو.

#### PASHTO ADOLESCENT ASSENT

# داو وان وګوهن په یو تخ واتي مطلع کې و تخ واتي مطلع کې ونتون

د **مطلعي عنوان:** د CoVID-9اپر اخ مرضهپر مالی د کهوال و مشومانی لپاره د هور<u>یمان</u>ی اولټولرهیز - احرماریشي زه کړې برنامچليمي کول او ارزونه: Empower

)د مه اجویق لپ اره کاورنی ک اوسال متعلیم څخمبه رد احسلريل وبرن امه (

اصلي څون وی ه ) دغه څوک چې دې څون ې مراوی تاري (: چای اروزنر ک MD MHS

(333 Cedar St, New Haven, CT)

د تهونشع ي ده: 860-930-1702

### ولى زلىت عم؟

- مورل متلس څخه غونوټه کوو چېپه څهرړي زهمطالعه کېږې خ ولئ.
  - مطلعمبه د دوبيهبرنامېس د ستمل وت جرب و کوري.
- دلبه دوه جلا مق ځېون کې شاو خو لی و ساعت و خت وغیسې ، د زو ل ه الريب وینون کې .

\_

- - ادفور مه د څه رن دوی ه مطاعې رض طات او سټملو ګډو زېه مطالع ه که ټووزي کو ي.
    - عهله دقتسر هېولولۍ او څومره وخت چې غواړ عپارې هې کاروی.
  - ه مهر ال يوکې کې حطال عې کار فيدلو څخه د هغه څهپه اړ مېوښتنې مېوښتنې چېټلاروپ رې نمېو هې د. ئ.
    - تىلىق كولى شى د مطاعى پ چون كى اوسى ا ەر وختىپ رىنى ئى بىيىنى ئى .
    - کامتسلوپ، مطالعه کی، در خالی، او کولی شی و روسته خال د ه نابلی کیرئ.
      - تىلىو ەر خت كولىشى مطلعمپوردى.
    - موربب سن بلس و مور اوپلار څخه مه و غواړو چې تلسوته اجازه دکړي په دې مطالعه کې دکړي.

## ولى دا مطلع ه لمته وړان يې يوي؟

موږل متىلسو څخه غوښته كوو چېپه څېړنى زهمطالعه كېبر خه ولځلئ ځكه چې**تىلسو اوستىلسوكورنى د ديې په بون امه** كې **برخه اځىئ**. موږ د **دغو مېلسولمړنى پانىټكې يو ئېپه بون امكې يې برخه خوستې ، اوش اوخوا 70تن م**ټول د دې مطاع يېبر خمشي يېر څو د دېپه اړمنور على ومات زه كړي چېبرن ام سټىلسو اوستېللو كورنۍ لېباره څه ده.

## مطلعه د څهشي په اړه ده؟

د دې مطاعې هدف د ه غوبرن امې ار زون ه ده چې سټملو کورن پې میک یېبر خه الحلي یې بار خه الحجيم و ي ، د EMPOWER په د د د کېږي .

## د مطلع په چانکه خه پیښشي؟

م برخه واځيئ ، چ پکې به او بېکول ، ده ن پرؤې شپېړول ، او دورغتى ا او هولى نې په اړه زدكړه ، او د 19-COVID غينى توب او اح لالكو په اړه زدكړه شامل وي.

## زو به څومره و ختالواړه په مطلع کی اس ی دم؟

تسلوبه د 2 زوم لی نېولرئ چېپه مري کېښاوخوا 1ساعت و خترېسي. دا د دېبرن امېسپېره دې کوم چېبه د دوه اوښيوپه اوږد کې د خضووي ګډون 3ساعته وي اوپه ولوۍ کې دڅلورو اوښي لپاره 1ساعتبه وم کې وي.

## د مطلعی حصملی خطرون کوم دی؟

تىلى و مكن د ئونى يېرىنىتى بوسىرە چې موږى ې غونىق كووى و خكىلى فىتىچىدە كېرئ مېدې مېزى چې مكن ئواب ھالى ي مركا ويى اد اچىلايلەق او اچىلايلەوپ، او فىكىركول او خىرى كولسخت وي بپە خطرون كې مكن سېرن امو څخ خەخوند انجىيتالى ان دخوشول مېش امل وي.

## څنګه به زه د مطلع په اړکوم نوي م هم ملي ومات زدک رم؟

مورب متملس و اوستملس ميال رينوت و ويلي که چهرې مورک و من و ي علومات زه کېړ و چې مکرنپ دېمطالعه ک بهبر خه الخهتال و په اړ دستملس فکربلي کېړي.

## څنګه مطلع کو لای شي ممکن لم یا نورو ځکو تیسته ورسوي؟

مطلاعه مکن نتاريټه ګنټه ورسوي متجيې لرلو له لملهپېوګرلم کې چېټلريوبه د دوييپېبرن له کېولرئ مپوشمول د نووي ليو د نووي ليوو اوتمړيزينو زهکېړه ، او د احمىلايګو او احمىلايګوپ اړه زهکېړه. مطلاع مشلىد دنوروخ لکوسره د EMPOWERبرن اممپه اړه د نوروپو محمد کې مرسټوکېړي او ه غوخ لک چې څخکه پېمبرن لمه کېښرخه ولح لي د دېپه اړه احمايل کېړي.

## اي الدبه زطلب ارده عسول عبن ولري؟

تعلى و اليخول لر عبيدي څخون ه كې لكښ توكې دى يى وازې لكښتون كې برن امېت متر رايه په ورتش امل دي.

## اي از مبه معاش وكرشمكه زه يه مطلع كىش املشم؟

تىلىوبىمپىدى څىن كېدىرخە الخهتالو لپارمتالى وركېرئ ستىلى كورنىبە د 25دالىرو دالى كارىتتىر لاس كېري. تىلىو مېرنېدى رىلىت كې مېلى كىد لەلمتالىيلو لپارە د دلت فىدرالىي بىانورومالىيلەوتىلە كولو مېرۇلورسى.مالى، ستىلىرو متالىيلە څخەن سرىك كىرى.

## زه نوركواختى ارون هارم؟

که تملسون، غواړئ د دې څيړنې پېرزخه و اوسئ متملسو ځينې نور لټ خپلې ه لرلۍ شي. تملي کوي شي:

- پتنه له مطاعې څخه د درملنې السو کول بتلسوکولی شي په MPOWER کې برخه واځی څومو یا
  څومړو لې چې تلوی یې غواړ ی کمان ه یلایت یا نه مطلح ته ادامه و کول لې پاره غورکوئ.
  - پېمالمېرنامه کېمېرخه ولځلئ.

## تىلى و زما مى وماتخنى خوندى ساتى؟

مورب سن ماره هغه عل ومات ت کړو چې محرم وي.

مونږب هې ې نوروس ره شوک کړو که تمال و موفل ق مهال ت کهال چې موږبلی د دلت رس و کړو ځکه چې د مټرده ۱۱۱لت د قرالون له مخې د لواالت ورته اړتا لري . د مڅال پ متوګه ، موږب ه و چله و ولی و که موږپ و شو چېتمال وی و مهل و چې ا ز او کس ته نی ان رس و ی.

ټول هغه چلومات چېټمل*ىوىېشو*ک کوئ هغمبه خوند*يک مچەپټارک ې* چېپسورډولري وسيلىلشي. موږبستىلىونوم ستىلىو ځويلونەسرە نىر مەنگىړو ، ئېر د هغېپه ځاىب، شېرنىنېشىمروكاروو.

کــله چې موږ د څۍړنېپيالې خپرووييله کښرراښين کــې د دېپه اړه غړېږو، موږب سټللونوم نو،ه کــاروو. کــه موږ غواړو چې ښټللونو وکاروو ، موږبه ل متللو څخه د اجازې غړښتن وکــړو.

موږ مکن سټمل وټه اړه عل ومات د ټالونځ ي څهري لپارهن ورو څه ړونځ و سره ممش وکټ کېړو کېر موږب سټمل ون و مېان نور شرن اخت و کورځ کېږي که د کومخالفي اجازې غوښتن و وکېږي که د و د د کومخالفي اجازې غوښتن و وکېږي د .

#### ای ا و بلی په دی مطلع کی ش امل شم؟

نه مپدې مطالعه کـ کهبر خه المحیت لهتمل ویپورې اړه لري بتملو کولی شئ او سنه و ولیملان که کمتمل و دم خهپو می برئ چې پهتمل و نه غواړئ په کېدې که تملل و نه غواړئ په کېدې کې که تملل و نه غواړئ کـ پې که تملل و نه غواړئ کـ پې که تملل و نه کولی شئ هم دا او س ه و وی لی کـ همتمل و نور نه غواړئ د دېبر خهشئ. کولی شئ هر و خت مطالع مپهرونک یې د دېبر خهشئ. څه پر ونځ کې ال هم ه غه چل و ماتوکاروي چې دم خه مېسټمل ویپه اړه ریالي کـ پري م کې له دې چې تمل و د مطاعې څه د دې پې تمل و د مطاعې څه دې پې تمک له دې چې تمل و د مطاعې څه دې پې تورشي م

ه څ فه ي پوللې به فه لري پوته ل دې چې د هغه څوپه اړ مپوکې وکې ئ چېتلري ې کو ئ سټللوپ وکې رهبه هغه الهرن ه بدل مرکې د ي چېتللوي ېټر لاره کو ي ي اغه ګټې چېتللوي ېې پان د ولت ر لاره کو ئ.

څېړورکۍ يې مکن تندل وپ مت څوق کې د بره الحیمتال و څخه ل چې کې ړيکه اړی ا و ب**یبه تندل و یس تندل وکورنۍ نور ن ه غواړ**ئ برخه واځی، تندل و ممکن هر وځتبرخ**ه خون نی** بویږدی.

## څ مکه و سنووتنی ولرم؟

مه بازيوكې د ور څخه د هر هغه څوه اړ مېونتون وكې ي چېتلارون و وبال دېپو يې رئ.

كەتىلىرو وروسىتەمپىينىتىنى، بولىرىن كەتىلىرو د مطاعېسىرەسىتىرىن ئىلىق كولىي شېھە كىي دىمطال عې مىرۇل لېكىتىرىت، پىدى شەھىرە 860- 1702-1702 زنگ وو ەئ.

## اجازه او واک وکول

ستملسو لهفقه کومه چې موړيبهې اوسستملسو اجازېسره مېتن کېړو ، دپله ګنتوه کوي چېتملسو دا د رضمت فور مه او وړل دېشو ي ځلومات اويمېدلي اوپويهدلي يې او دا چېتملسو مغلق پهلستېدې څېړړه کېښه اوسئ.

مو رب متلاوت د دي اجازه اي کمپلي چټو کړو.

#### PASHTO CHILD ASSENT

## 

سرلي ک: د Empower برنام يې وينتنې.

## ز مولي دل*ټىم*؟

موږلمتىلىو څخە غونيوتپە كىوو چېپىصوە څېړرنىزە مطالع، كىببىر خە ولجلىئ ئېكە چې موږ څە كىوو چېستىلىرو د احمىلايىلتو او احمىلايىلتەيپە اړەنور چلومات زەكىړو. مورتتىلىوتىپە مطلاعكى د گىدونيىلىنە دكىوو ئېكە چېتىللىوپىدېىدىي كىب پەMPOWER-يېبىر خەلجلىئ.

## دو يولي دامطالعه كوي؟

موړ غواړو د EMPOWERپمېرن امېوه شو او EMPOWER مکنېدل شي چې څګه تملسو د حولسو او احمل لويلتو په او فک رک و ئ

## زماس مبه څه کیږي؟

تىلىوب د دوبى پېمېرن لم كې د لويو لويولو پرځ مكولي فعالىتېن وترس و كولو ، او د COVID-19 خون يو بې اړ ه زده كې كېيېرخ ه ولحلئ. موږب لمتىلس څخه د زويې ه كېپونينې مېركېړو. موږب مېينينوت دو ه مظاف و تېون ه وكېړو. تىلل و مېن ورت پونينې دو ه ځله و او رئ.

## عى مطلعمبه زيان ورسوي؟

## عی مطل عمبه ز ماس ه مرست و کې ي؟

موږ لمهد لرو چې د MPOWERبرزلمه کـــېـــــر خه المچينټالب.مستملسو احربلايهاتو او احربلايهاتوسره مرسټوکـــړي ، ګـــر موږ ډاډهن.هــو چې داسېبه وښي.

## څه که و کومهپوښتن ولرم؟

تىلى كولىشكى، كومېپونىتىنى د مطاعېپ، اړه لىرى ھېۋىتى. كىمىلىن و روستىھى مېونىتىن مولىرى چېتىلىرى، اوسېپ، او فكىرن دىش كىورى مىلىق كولىش،ئې، دېشھىرە) 1702-930-86(بىلدىتىلغىوزوكىدى ئىلبىل ځل زما څخېونىتىن، وكېرى.

د دې او که يې آز مون يې وضري حاتب په http://www.ClinicalTrials.gov پې الکه څې ه چې د مې حده عااله و و لو او او الري بې د دې ه به بې اه که بې له ومات شامل ن ه و ي چېتل و پې ژني. حاکمتر په دی هې به پاڼک ي د د پالو لون ه زش امل و ي بتلو کول ي ش که د ه به په اړه و خت کې و ري.

## <u>لي از ماوال في نيدي اړميو عي دي؟</u>

دا څه ړڼ سټلسو مور اوپلارت متوضري حشوې او دوی و هال چېټلل وې پدونځولی شی بتلو کولی شئ مځې ل دې چې ل دې چې په کې چې پې کوکې ړ و کې ړئ دوی س ره دا خېرې و کې ئ

#### على ز مبطىدب مطالعه كى اوسم؟

تىلى و اېرى الى ئېدەمطالىخە كىمى اوسىئ. ئىڭوكىبەن اراض شىرى كەتىلى دان، غواړئ. كەتىلى ون، غواړ ئېدى څىز ، كىمى اوسىئ ،نوتىلى وبىلى دوىت، وولىلىت بىلىق كولى شىئ ەمدا اوس ەو وولى يى او وروست، شى فىكىرىبىكى كېرئ بېمىلى وپ ورى ارە لىرى.